CLINICAL TRIAL: NCT00000310
Title: Serotonin/Dopamine Antagonism of Cocaine Effect
Brief Title: Serotonin/Dopamine Antagonism of Cocaine Effect: 2 - 2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09330-2; R01-09330-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 1996-01

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
The purpose of this study is to evaluate use of risperidone with cocaine abusers. Study measures incorporate an appropriate integration of behavioral and neurobiological indices.

DETAILED DESCRIPTION:
Risperidone in low doses is compared with placebo in a 6-week randomized trial. Subjects also receive supportive counseling. Outcome measure include rating of behavior, mood, drug abuse, global function, and urine toxicology.

ELIGIBILITY:
Inclusion Criteria:

Cocaine abuse or dependence

Exclusion Criteria:

Dependence on other drugs. Major psychiatric illness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-01; Primary Completion 1996-03 (Actual); Study Completion 1996-03 (Actual)

PRIMARY OUTCOMES:
Urine toxicology for cocaine
Analog mood scales
POMS
EPS sx

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Price, M.D., Principal Investigator — Brown University
Locations (1):
- Brown University School of Medicine, Providence, Rhode Island, United States